CLINICAL TRIAL: NCT04995419
Title: A Single-arm, Open-label, Multi-center Phase 2 Study of Enfortumab Vedotin (ASG-22CE) in Chinese Subjects With Locally Advanced or Metastatic Urothelial Cancer Who Previously Received Platinum-containing Chemotherapy and PD 1/PD-L1 Inhibitor Therapy (EV-203)
Brief Title: A Study to Evaluate Enfortumab Vedotin (ASG-22CE) in Chinese Participants With Locally Advanced or Metastatic Urothelial Cancer Who Previously Received Platinum-containing Chemotherapy and Programmed Cell Death Protein-1 ( PD 1) / (Programmed Death Ligand-1 (PD-L1) Inhibitor Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7465-CL-1104; CTR20210922 (Registry Identifier: chinadrugtrials.org.cn)
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Urothelial Cancer
Keywords: Enfortumab Vedotin; PADCEV; ASG-22CE; Pharmacokinetics; Urothelial cancer
MeSH Terms: interventions — enfortumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Enfortumab Vedotin 1.25 mg/kg (Experimental): Participants received 1.25 milligrams per kilogram (mg/kg) of body weight enfortumab vedotin by intravenous (IV) infusion over approximately 30 minutes on days 1, 8 and 15 of every 28-day cycle. Participants received study treatment until radiological disease progression as determined per investigator assessment or other discontinuation criteria were met or upon study termination, or study completion, whichever occurred first. Participants who had intense PK Sampling were enrolled in PK Cohort.
  Interventions: Drug: Enfortumab vedotin

INTERVENTIONS:
Drug: Enfortumab vedotin — Intravenous Infusion
  Other Names: PADCEV, ASG-22CE

SUMMARY:
The purpose of this study was to determine the antitumor activity of enfortumab vedotin (EV) confirmed by the objective response rate (ORR).

This study also evaluated the effect of antibody-drug conjugate (ADC), total antibody (TAb) and monomethyl auristatin E (MMAE) in Chinese participants with locally advanced or metastatic urothelial cancer.

In addition, the study also evaluated the duration of response (DOR), disease control rate (DCR), progression-free survival (PFS), overall survival (OS), and immunogenicity determined by the incidence of antitherapeutic antibodies (ATA).

Safety and tolerability of EV in participants with locally advanced or metastatic urothelial cancer was also evaluated.

DETAILED DESCRIPTION:
This study comprised of a single group of participants who received one dose of enfortumab vedotin (EV) on Days 1, 8 and 15 of every 4-week (28 days) cycle. Participants continued on study treatment until discontinuation.

After treatment discontinuation, participant had an end of treatment (EOT) visit for a 30-day Safety Follow-up.

Participants to discontinue to treatment for reasons other than disease progression were followed for response assessments.

A Pharmacokinetic (PK) cohort was available at some study centers. Participants enrolled at the PK cohort site(s) had intense PK samples collected after single and repeated doses.

ELIGIBILITY:
Inclusion Criteria:

* Participant has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participant must have histologically or cytologically documented urothelial/transitional cell carcinoma of the bladder, renal pelvis, ureter or urethra. Other histologies including adenocarcinoma, squamous differentiation or mixed are eligible.
* Participant has locally advanced or metastatic disease that is not amenable to curative intent treatment. Participants must have measurable disease at baseline according to Response Evaluation Criteria in Solid Tumors (RECIST) ( Version 1.1). Lesions in a prior radiation field must have progressed subsequent to radiotherapy to be considered measurable.
* Participant must have received prior treatment with PD-1/PD-L1 inhibitor therapy in the locally advanced or metastatic urothelial cancer setting. Participants who received PD-1/PD-L1 therapy in the neoadjuvant/adjuvant setting and had recurrent or progressive disease either during therapy or within 3 months of therapy completion are eligible.
* Participant who received prior treatment with platinum-containing chemotherapy defined as those who received platinum in the neoadjuvant/adjuvant setting and had recurrent or progressive disease within 12 months of completion or received treatment with platinum in the locally advanced (defined as unresectable with curative intent) or metastatic setting.

  * Platinum based chemotherapy may include combination use with a PD-1 or PD-L1 inhibitor.
* Participant has the following baseline laboratory data. If a participant has received a recent blood transfusion or growth factor, the hematology tests must be obtained ≥7 days after any growth factor and ≥ 28 days after any blood transfusion.

  * absolute neutrophil count (ANC) ≥ 1.0 × 10^9/L
  * platelet count ≥ 100 × 10^9/L
  * hemoglobin ≥ 9 g/dL
  * serum total bilirubin (TBL) ≤ 1.5 × upper limit of normal (ULN) or ≤ 3 × ULN for participants with Gilbert's disease
  * creatinine clearance (CrCl) ≥ 30 mL/min as estimated per institutional standards or as measured by 24-hour urine collection (glomerular filtration rate [GFR] can also be used instead of CrCl).
  * alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN
* Female participant is not pregnant and at least one of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 6 months after the last dose of study treatment administration.
* Female participant must agree not to breastfeed starting at screening and throughout the study period and for at least 6 months after the last dose of study treatment administration.
* Female participant must not donate ova starting at first dose of study treatment and throughout the study period and for 6 months after the last dose of study treatment administration.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for 6 months after the last dose of study treatment administration.
* Male participant must not donate sperm during the treatment period and for 6 months after the last dose of study treatment administration.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 6 months after the last dose of study treatment administration.
* Participant agrees not to participate in another interventional study while receiving study treatment in the present study.
* Participant must have had progression or recurrence of urothelial cancer during or following receipt of most recent therapy.
* Participant must have an anticipated life expectancy of ≥ 3 months.

Exclusion Criteria:

* Participant has preexisting sensory or motor neuropathy Grade ≥ 2.
* Participant has active central nervous system (CNS) metastases. Participants with treated CNS metastases are permitted on study if all the following are true:

  * CNS metastases have been clinically stable for ≥ 6 weeks prior to screening.
  * If requiring steroid treatment for CNS metastases, the participant is on a stable dose ≤ 20 mg/day of prednisone or equivalent for ≥ 2 weeks.
  * Baseline imaging scans show no evidence of new or enlarged brain metastasis.
  * Participant does not have leptomeningeal disease.
* Participant has ongoing clinically significant toxicity (Grade 2 or higher with the exception of alopecia) associated with prior treatment (including systemic therapy, radiotherapy or surgery).
* Participant with ongoing ≥ Grade 3 immunotherapy-related hypothyroidism or panhypopituitarism is excluded. Participant with ongoing immunotherapy-related colitis, uveitis, myocarditis or pneumonitis, or participants with other immunotherapy-related AEs requiring high doses of steroids (> 20 mg/day of prednisone or equivalent), is excluded. Participant with ≤ Grade 2 immunotherapy-related hypothyroidism or panhypopituitarism may be enrolled when well-maintained/controlled on a stable dose of hormone replacement therapy (if indicated).
* Participant has a history of uncontrolled diabetes mellitus within 3 months before the first dose of study treatment. Uncontrolled diabetes is defined as hemoglobin A1c (HbA1c) ≥ 8 percent or HbA1c between 7 percent and < 8 percent with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained.
* Participant has prior treatment with enfortumab vedotin or other monomethyl auristatin E (MMAE)-based antibody-drug conjugate (ADCs).
* Participant has a second malignancy diagnosed within 3 years before first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Participants with non-melanoma skin cancer, localized prostate cancer treated with curative intent with no evidence of progression, low-risk or very low-risk (per standard guidelines) localized prostate cancer under active surveillance/watchful waiting without intent to treat, or carcinoma in situ of any type (if complete resection was performed) are allowed.
* Participant is currently receiving systemic antimicrobial treatment for viral, bacterial or fungal infection at the time of first dose of study treatment. Routine antimicrobial prophylaxis is permitted.
* Participants with a positive hepatitis B surface antigen and/or anti-hepatitis B core antibody and a negative polymerase chain reaction (PCR) assay at baseline should receive appropriate antiviral prophylaxis or regular surveillance monitoring as per local or institutional guidelines.
* Active hepatitis C infection or known human immunodeficiency virus (HIV) infection. Participant who have been treated for hepatitis C infection are permitted if they have documented sustained virologic response of ≥ 12 weeks.
* Participant has documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction or cardiac symptoms (including congestive heart failure) consistent with New York Heart Association Class III-IV within 6 months prior to the first dose of study drug.
* Participant had major surgery within 2 weeks or radiotherapy, chemotherapy, biologics, investigational agents, and/or antitumor treatment with immunotherapy that is not completed 2 weeks prior to first dose of study drug. Toxicities from these therapies must have resolved or adequately stabilized before starting study treatment.
* Participant has known hypersensitivity to enfortumab vedotin or to any excipient contained in the drug formulation of enfortumab vedotin (including histidine, trehalose dihydrate and polysorbate 20) or participant has known hypersensitivity to biopharmaceuticals produced in CHO cells.
* Participant has known active keratitis or corneal ulcerations. Participant with superficial punctate keratitis is allowed if the disorder is being adequately treated.
* Participant has any condition which makes the participant unsuitable for study participation.
* Uncontrolled tumor-related bone pain or impending spinal cord compression. Participant requiring pain medication must be on a stable regimen for at least 2 weeks at the time of first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2025-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Science Manager, Study Director — Astellas Pharma China, Inc.
Locations (7):
- China (7):
  - Site CN86001, Beijing
  - Site CN86009, Changsha
  - Site CN86002, Guangzhou
  - Site CN86006, Hangzhou
  - Site CN86007, Nanjing
  - Site CN86004, Shanghai
  - Site CN86003, Wuhan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Li S, Shi Y, Dong H, Guo H, Xie Y, Sun Z, Zhang X, Kim E, Zhang J, Li Y, Xu C, Kadeerbai H, Lee S, Gorla S, Guo J, Sheng X. Phase 2 Trial of Enfortumab Vedotin in Patients With Previously Treated Locally Advanced or Metastatic Urothelial Carcinoma in China. Cancer Med. 2024 Nov;13(21):e70368. doi: 10.1002/cam4.70368. PMID 39530574

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult Chinese participants with locally advanced or metastatic urothelial cancer (mUC) who had received a platinum-containing chemotherapy and programmed cell death protein-1 (PD-1) or programmed death-ligand 1 (PD-L1) inhibitors.
Pre-assignment Details: Participants who met inclusion criteria and none of the exclusion criteria were enrolled.
Groups:
- Enfortumab Vedotin 1.25 mg/kg: Participants received 1.25 milligrams per kilogram (mg/kg) of body weight enfortumab vedotin by intravenous (IV) infusion over approximately 30 minutes on days 1, 8 and 15 of every 28-day cycle. Participants received study treatment until radiological disease progression as determined per investigator assessment or other discontinuation criteria were met or upon study termination, or study completion, whichever occurred first.
Period: Overall Study
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Started | 40
Completed | 0
Not Completed | 40
Not completed — Withdrawal by Subject | 3
Not completed — Progressive Disease | 19
Not completed — Adverse Event | 2
Not completed — Ongoing | 16

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were enrolled and received any amount of study drug in the study.
Groups:
- Enfortumab Vedotin 1.25 mg/kg: Participants received 1.25 mg/kg of body weight enfortumab vedotin by IV infusion over approximately 30 minutes on days 1, 8 and 15 of every 28-day cycle. Participants received study treatment until radiological disease progression as determined per investigator assessment or other discontinuation criteria were met or upon study termination, or study completion, whichever occurred first.
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 40
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Per Response Evaluation Criteria in Solid Tumors V1.1 (RECIST V1.1)
Description: ORR was defined as the percentage of participants with best overall response (BOR) as complete response (CR) or partial response (PR) based on the RECIST v1.1. CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
Time Frame: From first dose up to progressive disease or death (maximum duration: 9.33 months)
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 40
percentage of participants | 37.5 [22.7 to 54.2]

2. Primary Outcome: Pharmacokinetics (PK) of Antibody-Drug Conjugate (ADC), Total Antibody (TAb), in Serum: Maximum Concentration (Cmax) at Cycle 1 Day 1
Description: Cmax was derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 1: pre-dose, end of infusion (EOI), 2 hour, 4 hour post-dose (each cycle = 28 days)
Population: Pharmacokinetic Analysis Set (PKAS) included all participants in the PK cohort who had received at least 3 of 4 doses up through Cycle 2 Day 1, and had at least 5 blood samples collected and assayed for measurement of ADC, TAb or unconjugated MMAE serum/plasma concentrations to determine at least 1 PK parameter.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (ug/mL)
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 13
micrograms per milliliter (ug/mL)
  ADC | 28.1 (4.52)
  TAb | 31.7 (5.73)

3. Primary Outcome: PK of Monomethyl Auristatin E (MMAE) in Serum: Maximum Concentration (Cmax) at Cycle 1 Day 1
Description: Cmax was derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 1: pre-dose, end of infusion (EOI), 2 hour, 4 hour post-dose (each cycle = 28 days)
Population: PKAS population.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 13
nanograms per milliliter (ng/mL) | 3.33 (1.74)

4. Primary Outcome: PK of ADC, TAb in Serum: Maximum Concentration (Cmax) at Cycle 1 Day 15
Description: Cmax was derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 15: pre-dose, EOI, 2 hour, 4 hour post-dose (each cycle = 28 days)
Population: PKAS population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 10
ug/mL
  ADC | 27.6 (4.01)
  TAb | 34.4 (4.64)

5. Primary Outcome: PK of MMAE in Serum: Maximum Concentration (Cmax) at Cycle 1 Day 15
Description: Cmax was derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 15: pre-dose, EOI, 2 hour, 4 hour post-dose (each cycle = 28 days)
Population: PKAS population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 10
ng/mL | 4.49 (3.58)

6. Primary Outcome: PK of ADC , TAb in Serum: Trough Concentration (Ctrough) at Cycle 1 Day 1
Description: As per planned analysis, if more than 50% of PK concentrations were below the limit of quantification (i.e 0) at a given time point, standard deviation was not reported.
Time Frame: Cycle 1 Day 1: pre-dose
Population: PKAS population.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 13
ug/mL
  ADC | 0 (NA) — Standard Deviation was not reported in summary statistics because more than 50% of ADC concentrations at pre-dose were 0.
  TAb | 0 (NA) — Standard Deviation was not reported in summary statistics because more than 50% of TAb concentrations at pre-dose were 0.

7. Primary Outcome: PK of MMAE in Serum: Trough Concentration (Ctrough) at Cycle 1 Day 1
Description: as for outcome 6
Time Frame: Cycle 1 Day 1: pre-dose
Population: PKAS population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 13
ng/mL | 0 (NA) — Standard Deviation was not reported in summary statistics because more than 50% of MMAE concentrations at pre-dose were 0.

8. Primary Outcome: PK of ADC, TAb in Serum: Trough Concentration (Ctrough) at Cycle 1 Day 15
Description: Ctrough was derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 15: pre-dose
Population: PKAS population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 12
ug/mL
  ADC | 1020 (410)
  TAb | 4620 (1590)

9. Primary Outcome: PK of MMAE in Serum: Trough Concentration (Ctrough) at Cycle 1 Day 15
Description: Ctrough was derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 15: pre-dose
Population: PKAS population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 12
picograms per milliliter (pg/mL) | 1880 (1680)

10. Primary Outcome: PK of ADC, TAb, MMAE in Serum: Time to Maximum Concentration (Tmax) at Cycle 1 Day 1
Description: Tmax was derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 1: pre-dose, EOI, 2 hour, 4 hour post-dose (each cycle = 28 days)
Population: PKAS population.
Measure: Median (Full Range); unit: days
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 13
days
  ADC | 0.0340 [0.0278 to 0.0917]
  TAb | 0.0340 [0.0243 to 1.89]
  MMAE | 2.00 [1.87 to 2.93]

11. Primary Outcome: PK of ADC, TAb, MMAE in Serum: Time to Maximum Concentration (Tmax) at Cycle 1 Day 15
Description: Tmax was derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 15: pre-dose, EOI, 2 hour, 4 hour post-dose (each cycle = 28 days)
Population: PKAS population with available data were analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 10
days
  ADC | 0.0337 [0.0257 to 0.0805]
  TAb | 0.0337 [0.0278 to 0.0854]
  MMAE | 1.93 [0.858 to 2.92]

12. Primary Outcome: PK of ADC, TAb, MMAE in Serum: Area Under Concentration-time Curve From 0 to Day 28 (AUC0-28d) at Cycle 1 Day 1
Description: AUC0-28d was derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 1: pre-dose, EOI, 2 hour, 4 hour post-dose (each cycle = 28 days)
Population: Per protocol, data for AUC0-28d was planned to be calculated using non-compartment analysis (NCA) only if data permits, therefore AUC 0-28d was removed from the planned analysis in SAP.
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 0

13. Primary Outcome: PK of ADC, TAb, MMAE in Serum: Area Under Concentration-time Curve From 0 to Day 28 (AUC0-28d) at Cycle 1 Day 15
Description: AUC0-28d was derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 15: pre-dose, EOI, 2 hour, 4 hour post-dose (each cycle = 28 days)
Population: as for outcome 12
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 0

14. Primary Outcome: PK of ADC, TAb in Serum: Area Under Concentration-time Curve From 0 to Day 7 (AUC0-7d) at Cycle 1 Day 1
Description: AUC0-7d was derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 1 : pre-dose, EOI, 2 hour, 4 hour post-dose (each cycle = 28 days)
Population: PKAS population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 12
day*ug/mL
  ADC | 32.4 (6.24)
  TAb | 77.4 (17.3)

15. Primary Outcome: PK of MMAE in Serum: Area Under Concentration-time Curve From 0 to Day 7 (AUC0-7d) at Cycle 1 Day 1
Description: AUC0-7d was derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 1 : pre-dose, EOI, 2 hour, 4 hour post-dose (each cycle = 28 days)
Population: PKAS population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 12
day*ng/mL | 16.9 (9.21)

16. Primary Outcome: PK of ADC, TAb in Serum: Area Under Concentration-time Curve From 0 to Day 7 (AUC0-7d) at Cycle 1 Day 15
Description: AUC0-7d was derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 15: pre-dose, EOI, 2 hour, 4 hour post-dose (each cycle = 28 days)
Population: PKAS population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 10
day*ug/mL
  ADC | 36.5 (7.93)
  TAb | 94.7 (15.7)

17. Primary Outcome: PK of MMAE in Serum: Area Under Concentration-time Curve From 0 to Day 7 (AUC0-7d) at Cycle 1 Day 15
Description: AUC0-7d was derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 15: pre-dose, EOI, 2 hour, 4 hour post-dose (each cycle = 28 days)
Population: PKAS population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 10
day*ng/mL | 23.3 (16.4)

18. Primary Outcome: PK of ADC, TAb, MMAE in Plasma: Accumulation Ratio of Cmax (RacCmax)
Description: Accumulation ratio is the ratio of Cmax after the dosing interval (Cycle 1 Day 15) divided by Cmax after the first dosing interval (Cycle 1 Day 1).
Time Frame: Cycle 1 Day 15: pre-dose, EOI, 2 hour, 4 hour post-dose (each cycle = 28 days)
Population: PKAS population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 10
ratio
  ADC | 1.03 (0.150)
  TAb | 1.13 (0.137)
  MMAE | 1.28 (0.499)

19. Primary Outcome: PK of ADC, TAb, MMAE in Serum: Accumulation Ratio of AUC0-7d ( RacAUC0-7d)
Description: RacAUC0-7d was calculated using AUC0-7d and derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 15: pre-dose, EOI, 2 hour, 4 hour post-dose (each cycle = 28 days)
Population: PKAS population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 10
ratio
  ADC | 1.20 (0.228)
  TAb | 1.29 (0.208)
  MMAE | 1.32 (0.486)

20. Primary Outcome: PK of ADC, TAb, MMAE in Serum: Terminal Elimination Half-life (t1/2)
Description: t1/2 was derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 15: pre-dose, EOI, 2 hour, 4 hour post-dose (each cycle = 28 days)
Population: PKAS population with available data were analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 10
days
  ADC | 2.81 [2.28 to 3.70]
  TAb | 3.82 [3.11 to 5.49]
  MMAE: number analyzed (Participants) | 9
  MMAE | 3.12 [2.83 to 3.82]

21. Primary Outcome: PK of ADC, TAb, MMAE in Serum: Systemic Clearance (CL)
Description: CL was derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 15: pre-dose, EOI, 2 hour, 4 hour post-dose (each cycle = 28 days)
Population: PKAS population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Liters/hour (L/hr)
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 10
Liters/hour (L/hr)
  ADC | 0.104 (0.0239)
  TAb | 0.0396 (0.00847)
  MMAE | 196 (76.2)

22. Primary Outcome: PK of ADC, TAb, MMAE in Serum: Volume of Distribution at Steady State (Vss)
Description: Vss was derived from the PK blood samples collected.
Time Frame: Cycle 1 Day 15: pre-dose, EOI, 2 hour, 4 hour post-dose (each cycle = 28 days)
Population: PKAS population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 10
Liters
  ADC | 7.13 (1.39)
  TAb | 4.97 (1.27)
  MMAE: number analyzed (Participants) | 9
  MMAE | 28900 (10800)

23. Secondary Outcome: Duration of Response (DOR) as Per RECIST V1.1 Per IRC
Description: DOR: time from the date of the first CR/PR (whichever is first recorded) that was subsequently confirmed as assessed by IRC to the date of documented progressive disease. or death due to any cause whichever occurred first. CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters. Progressive Disease:>= 20% increase in sum of diameters of target lesions taking as reference the smallest sum, and sum must also demonstrate an absolute increase of >= 5 mm. Appearance of 1 or more new lesions is also considered progression.
Time Frame: From date of the first CR/PR up to progressive disease or death (maximum duration: 9.33 months)
Population: FAS population with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 15
months | NA [2.04 to NA] — Due to low number of events, median and upper limit of CI was not estimable.

24. Secondary Outcome: Duration of Response (DOR) as Per RECIST V1.1 Per Investigator's Assessment
Description: DOR: time from the date of the first CR/PR (whichever is first recorded) that was subsequently confirmed as assessed by Investigator's Assesment to the date of documented progressive disease or death due to any cause whichever occurred first. CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters. Progressive disease:>= 20% increase in sum of diameters of target lesions taking as reference the smallest sum, and sum must also demonstrate an absolute increase of >= 5 mm. Appearance of 1 or more new lesions is also considered progression.
Time Frame: From date of the first CR/PR up to progressive disease or death (maximum duration: 9.33 months)
Population: FAS population with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 17
months | NA [2.04 to NA] — Due to low number of events, median and upper limit of CI was not estimable.

25. Secondary Outcome: Objective Response Rate (ORR) as Per Investigator Assessment
Description: ORR was defined as the percentage of participants with BOR as CR or PR based on the RECIST v1.1 as per investigator's assesment. CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
Time Frame: From first dose up to progressive disease or death (maximum duration: 9.33 months)
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 40
percentage of participants | 42.5 [27.0 to 59.1]

26. Secondary Outcome: Disease Control Rate (DCR) as Per RECIST V1.1 Per IRC
Description: DCR: percentage of participants with a CR, PR or SD based on RECIST v1.1 as assessed by IRC. CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters. SD was defined as neither sufficient decrease to qualify for PR nor sufficient increase to qualify for progressive disease taking as reference the smallest sum of diameters while on study drug. Progressive disease:>= 20% increase in sum of diameters of target lesions taking as reference the smallest sum, and sum must also demonstrate an absolute increase of >= 5 mm. Appearance of 1 or more new lesions is also considered progression.
Time Frame: From first dose up to progressive disease or death (maximum duration: 9.33 months)
Population: FAS population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 40
percentage of participants | 72.5 [56.1 to 85.4]

27. Secondary Outcome: Disease Control Rate (DCR) as Per RECIST V1.1 Per Investigator's Assesment
Description: DCR: percentage of participants with a CR, PR or SD based on RECIST v1.1 as assessed by investigator's assessment. CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters. SD was defined as neither sufficient decrease to qualify for PR nor sufficient increase to qualify for progressive disease taking as reference the smallest sum of diameters while on study drug. Progressive disease:>= 20% increase in sum of diameters of target lesions taking as reference the smallest sum, and sum must also demonstrate an absolute increase of >= 5 mm. Appearance of 1 or more new lesions is also considered progression.
Time Frame: From first dose up to progressive disease or death (maximum duration: 9.33 months)
Population: FAS population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 40
percentage of participants | 82.5 [67.2 to 92.7]

28. Secondary Outcome: Progression Free-Survival Per RECIST V1.1 Per IRC
Description: PFS: time from first dose of the study drug until date of documented radiological disease progression per IRC based on RECIST V1.1, or until death due to any cause, whichever occurred first. Progressive disease: >= 20% increase in sum of diameters of target lesions taking as reference the smallest sum, and sum must also demonstrate an absolute increase of >= 5 mm. Appearance of 1 or more new lesions is also considered progression. A participant who neither progressed nor died was censored at date of last radiological assessment (RA)/ date of randomization if no post-baseline RA was available. Participants who received any further anticancer therapy (ACT) for disease before radiological progression was censored at date of last RA before ACT started and participants who had PD/death after >=2 missed RAs were censored at last RA prior to 2 or more missed RAs. Kaplan-Meier estimates was used.
Time Frame: From first dose up to progressive disease or death (maximum duration: 9.33 months)
Population: FAS population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 40
months | 4.67 [3.65 to 5.62]

29. Secondary Outcome: Progression Free-Survival Per RECIST V1.1 Per Investigator's Assessment
Description: PFS: time from first dose of the study drug until date of documented radiological disease progression per investigator based on RECIST V1.1, or until death due to any cause, whichever occurred first. Progressive disease: >= 20% increase in sum of diameters of target lesions taking as reference the smallest sum, and sum must also demonstrate an absolute increase of >= 5 mm. Appearance of 1 or more new lesions is also considered progression. A participant who neither progressed nor died was censored at date of last RA/ date of randomization if no post-baseline RA was available. Participants who received any further ACT for disease before radiological progression was censored at date of last RA before ACT started and participants who had progressive disease/death after >=2 missed RAs were censored at last RA prior to 2 or more missed RAs. Kaplan-Meier estimates was used.
Time Frame: From first dose up to progressive disease or death (maximum duration: 9.33 months)
Population: FAS population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 40
months | 4.24 [3.75 to 7.20]

30. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first dose of the study drug until the documented date of death from any cause. OS was analyzed using Kaplan-Meier estimates. Participants who were still alive at the time of data cutoff date were to be censored at the last known alive date or at the data cutoff date, whichever was earlier.
Time Frame: From first dose up to death (maximum duration: 9.33 months)
Population: FAS population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 40
months | NA [6.74 to NA] — Due to low number of events, median and upper limit of CI was not estimable.

31. Secondary Outcome: Number of Participants With Antitherapeutic Antibodies (ATA)
Description: Number of participants with ATA were reported.
Time Frame: From first dose until 9.33 months
Population: FAS population with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 38
Participants
  Baseline Negative, Negative post-baseline | 37
  Baseline Negative, Positive post-baseline | 0
  Baseline Positive, Negative post-baseline | 1
  Baseline Positive, Positive post-baseline | 0

32. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An AE is any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. TEAE is defined as an adverse event observed after starting administration of the study drug and within 30 days after taking the last dose of study drug.
Time Frame: Baseline up to 9.33 months
Population: Safety analysis set (SAF) included all participants who were enrolled and received any amount of study drug in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 40
Participants | 40

33. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)
Description: ECOG performance status was measured on an 6 point scale. 0-Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5. Dead. Number of participants with ECOG PS was reported."
Time Frame: End of Treatment (Baseline up to 9.33 months)
Population: SAF population
Measure: Count of Participants; unit: Participants
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
Number analyzed (Participants) | 40
Participants
  ECOG PS= 0 | 2
  ECOG PS= 1 | 8
  ECOG PS= 2 | 1
  ECOG PS= 3 | 1
  ECOG PS= 4 | 0
  ECOG PS= 5 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 9.33 months
Description: SAF
Arm/Group | Enfortumab Vedotin 1.25 mg/kg
All-Cause Mortality (participants affected / at risk) | 10/40
Serious Adverse Events (participants affected / at risk) | 18/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enfortumab Vedotin 1.25 mg/kg (N=40)
Leukopenia (Blood and lymphatic system disorders) | 2 (5)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (2)
Cataract (Eye disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 5 (6)
Respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 (2)
Drug eruption (Skin and subcutaneous tissue disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)
Deep vein thrombosis (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enfortumab Vedotin 1.25 mg/kg (N=40)
Anaemia (Blood and lymphatic system disorders) | 28 (81)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 4 (6)
Dry eye (Eye disorders) | 3 (3)
Eye discharge (Eye disorders) | 5 (5)
Vision blurred (Eye disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 19 (25)
Diarrhoea (Gastrointestinal disorders) | 19 (31)
Dyspepsia (Gastrointestinal disorders) | 7 (10)
Dysphagia (Gastrointestinal disorders) | 6 (10)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (5)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 20 (39)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 12 (17)
Asthenia (General disorders) | 4 (4)
Fatigue (General disorders) | 10 (31)
Malaise (General disorders) | 6 (7)
Oedema peripheral (General disorders) | 7 (15)
Pyrexia (General disorders) | 14 (17)
Herpes dermatitis (Infections and infestations) | 2 (2)
Herpes virus infection (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 3 (4)
Skin infection (Infections and infestations) | 6 (8)
Urinary tract infection (Infections and infestations) | 3 (3)
Alanine aminotransferase increased (Investigations) | 18 (30)
Aspartate aminotransferase increased (Investigations) | 26 (43)
Bilirubin conjugated increased (Investigations) | 2 (8)
Blood bilirubin increased (Investigations) | 4 (18)
Blood bilirubin unconjugated increased (Investigations) | 2 (3)
Blood creatinine increased (Investigations) | 5 (7)
Blood glucose increased (Investigations) | 4 (5)
Blood lactate dehydrogenase increased (Investigations) | 2 (3)
Blood triglycerides increased (Investigations) | 2 (3)
Gamma-glutamyltransferase increased (Investigations) | 3 (5)
Glycosylated haemoglobin increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 3 (6)
Neutrophil count decreased (Investigations) | 19 (36)
Occult blood positive (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 9 (22)
Weight decreased (Investigations) | 10 (17)
White blood cell count decreased (Investigations) | 16 (43)
Decreased appetite (Metabolism and nutrition disorders) | 26 (46)
Hypercalcaemia (Metabolism and nutrition disorders) | 5 (20)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 20 (57)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 (17)
Hyperuricaemia (Metabolism and nutrition disorders) | 11 (24)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (22)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (22)
Hypochloraemia (Metabolism and nutrition disorders) | 5 (9)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 15 (28)
Hyponatraemia (Metabolism and nutrition disorders) | 13 (35)
Hypophosphataemia (Metabolism and nutrition disorders) | 7 (14)
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 10 (21)
Hypoaesthesia (Nervous system disorders) | 6 (7)
Neuropathy peripheral (Nervous system disorders) | 8 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 8 (15)
Dysuria (Renal and urinary disorders) | 3 (3)
Haematuria (Renal and urinary disorders) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (12)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (17)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Drug eruption (Skin and subcutaneous tissue disorders) | 4 (8)
Eczema (Skin and subcutaneous tissue disorders) | 3 (5)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Papule (Skin and subcutaneous tissue disorders) | 5 (5)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (27)
Rash (Skin and subcutaneous tissue disorders) | 17 (56)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (13)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 5 (5)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (5)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT04995419/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT04995419/SAP_001.pdf